CLINICAL TRIAL: NCT04119115
Title: Integrated Radiographic and Metabolomics Risk Assessment in Patients With Interstitial Lung Diseases
Acronym: IRM-ILD
Status: Terminated | Type: Observational
Why Stopped: Lack of resources and funding
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Girish B. Nair, MD, Pulmonary Medicine Physician, Corewell Health East
Other Study IDs: 2019-241
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Lung Diseases, Interstitial; Pulmonary Fibrosis
Keywords: lung disease; pulmonary fibrosis; precision medicine; metabolomics
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis; Lung Diseases | interventions — Phytoalexins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Interstitial Lung Disease (ILD): CT-V and metabolite analysis of breath and serum at baseline
  Interventions: Device: CT-V; Other: Metabolites
- COPD/Emphysema: Age-matched control: CT-V and metabolite analysis of breath and serum at baseline
  Interventions: Device: CT-V; Other: Metabolites
- Healthy Volunteers: Age-matched + /- 10 yrs controls: Metabolite analysis of breath and serum at baseline
  Interventions: Other: Metabolites

INTERVENTIONS:
Device: CT-V — CT-V is a newer computed tomography scan which is more comprehensive and tracks movement of the lungs.
  Other Names: Quantitative lung function imaging and lung compliance imaging
  Groups: COPD/Emphysema: Age-matched control; Interstitial Lung Disease (ILD)
Other: Metabolites — Metabolites are compounds which can be measured in biospecimens and may indicate a disease or biological process.

SUMMARY:
The purpose of this study is to find out if combining a state-of-the-art form imaging modality with metabolomics in different types of Interstitial Lung Diseases (ILD) patients compared to controls with chronic obstructive pulmonary disorder (COPD)/emphysema and healthy controls will be a better predictor of disease progression. ILD's are a group of chronic, progressive lung diseases. The most common ILD is idiopathic pulmonary fibrosis (IPF). Metabolomics provides a "snapshot" in time of all metabolites present in a biological sample. The imaging procedure should take approximately 20 minutes. All study related collections of samples will be done in a single visit if possible. There are no direct benefits to participants. This is not a treatment study.

DETAILED DESCRIPTION:
Interstitial lung diseases (ILD) are a group of chronic, progressive lung disorders. The most common ILD is idiopathic pulmonary fibrosis (IPF) with an average survival ranging between 2.5-5 years after diagnosis. The term pulmonary fibrosis means scarring of the lung tissue and is the cause of worsening shortness of breath. IPF can frequently affect the tissue between the air sacs in the lung called the interstitium and many other areas in lung (blood vessels and air passage ways). Earlier diagnosis of ILD is a prerequisite for better long-term outcomes. However, disease detection and assessment of progression are reliant on many varying host and environmental influences. As a result, patients with ILD are often misdiagnosed early in the disease process. Moreover, patients diagnosed with ILD have different disease courses and predicting which patient is at risk of progression is a challenging problem. Many personalized medicine approaches are being developed but there is a lack of available biomarkers in clinical practice. Biomarkers comes from a new experimental technique called metabolomics which is becoming widely used in medicine and biology for studying living organisms. The method measures the levels of large numbers of naturally occurring small molecules (called metabolites) that are present in the blood, saliva, breath and tissues. The pattern, or fingerprint, of metabolites in human samples can be used to learn about the health of an organism and perhaps allow physicians to diagnose, treat, and follow the progress of specific diseases. Clinical and functional models lack predictive ability to detect patients at risk of disease progression. Thus, there is an urgent need to develop accurate prediction models for disease diagnosis and assess treatment effects.

CT-derived ventilation (CT-V) imaging includes quantitative lung function imaging and lung compliance imaging. CT-V is a newer image processing based technique that uses mathematical modeling and scientific computing to gather changes in lung tissue volumes during the breathing cycle. Beaumont is currently using CT-V for radiotherapy planning. CT-V produces a full 3D map of ventilation/breathing, has better image resolution, provides pertinent measurable imaging information, and does not require a contrast agent. Thus, high-resolution anatomical and functional information can be derived using CT-V.

To better understand the functional and radiographic changes seen in patients with ILD, there is a need to further examine the downstream changes occurring at the level of proteins and metabolites. Metabolomics provides a "snapshot" in time of all metabolites present in a biological sample. Proteins alone or integrated with other systems, is a particularly informative tool for understanding disease biology in ILD patients.Using an untargeted metabolomics platform and profiling serum and breathe from the patients will determine if additional or more robust biomarkers of disease can be identified and, in conjunction with the assessment of regional ventilation differences through CT-V, will provide a better insight into disease process and further help with accurate prognostication.

Participants who have consented for the study and have meet all the inclusion criteria and none of the exclusion criteria will have one full inspiration and expiration CT, and two 4D-CT scans under two different pressures (5 and 10 cm water), except for healthy volunteers. They will have their breath profiled using Owlstone platform and serum collected for metabolomics testing within one week period. Participants will be asked to refrain from smoking one day prior to the study date. All study related sampling will be done in a single visit if possible and if not possible all study procedures and samples will be collected within a one week period.

Disease progression will be assessed using chart review over the next 24 months to assess standard of care pulmonary function evaluation and corresponding CT features respiratory hospitalizations and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years of age
* Patients with a PFT-Pulmonary function test </=3 month plus seven days
* Patients with idiopathic pulmonary fibrosis (IPF), or
* Patients with interstitial lung disease (ILD) other than IPF, or
* Patients with chronic obstructive pulmonary disease COPD/emphysema based on Principal's Investigator's assessment/review, or
* Control subject, someone without a diagnosis of above and deemed and "healthy control" by the PI.

COPD/emphysema and control subjects will be age matched +/-10 years to the ILD subjects.

Exclusion Criteria:

* Patients less than 18 years of age
* Patients with active malignancy in past one year, except for basal and squamous cell skin cancer
* Patients without a PFT-Pulmonary function test </=3 month plus seven days
* Pregnant females
* Cognitive impairment and unable to follow directions, per PI discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pulmonary outpatient clinic and interstitial lung disease clinic at Beaumont Hospital, Royal Oak
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Quantitative image lung function | baseline
  CT-V scores between inhalation and exhalation will be calculated at a voxel level on each lung using the "Integrated Jacobian Formulation" (IJV) CT-V method in patients with IPF, non-IPF ILD and COPD/emphysema patients. Several factors, including the volume of identified "cold spots" (areas with decreased ventilation), total ventilation (the integral of CT-V image over the whole lung), and texture analytics (local means, variances, etc.) will be used to define a CT-V pulmonary function metric. This measure is reported in liters with lower numbers indicating reduced lung function.
Forced Vital Capacity baseline | baseline
  Maximum volume exhaled in liters measured on a spirometer at baseline

SECONDARY OUTCOMES:
Untargeted Metabolic profile of breath | baseline
  Identity and mean relative concentration of the most discriminating 10 volatile organic compounds identified by Owlstone untargeted metabolomic analysis, using mass spectrometry coupled with liquid and/or gas chromatography and robust bioinformatics, and normalized to controls. A value greater than one indicates increased concentration of the compound, and a value less than one indicates decreased concentration of the compound relative to the concentration in controls.
Untargeted Metabolic profile of Serum | baseline
  Identity and mean relative concentration of the most discriminating 10 compounds identified by untargeted metabolomic analysis of serum using mass spectrometry coupled with liquid and/or gas chromatography and robust bioinformatics and normalized to controls. A value greater than one indicates increased concentration of the compound, and a value less than one indicates decreased concentration of the compound relative to the concentration in controls.

CONTACTS AND LOCATIONS:
Overall Officials: Girish B Nair, MD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Health, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No